CLINICAL TRIAL: NCT05907668
Title: IMVT-1401-2501: A Proof-of-Concept, Open-label Study to Assess the Safety and Efficacy of Batoclimab in Participants With Graves' Disease (GD)
Brief Title: A Proof-of-Concept Study to Assess Batoclimab in Participants With Graves' Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMVT-1401-2501
Record Dates: First submitted 2023-05-15; First posted 2023-06-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Graves Disease
Keywords: Graves' Disease; IMVT-1401; Batoclimab; Hyperthyroidism
MeSH Terms: conditions — Graves Disease; Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Batoclimab (Experimental): Participants will receive batoclimab 680 milligrams (mg) subcutaneously (SC) weekly (QW) injection for 12 weeks followed by 340 mg SC QW for 12 weeks.
  Interventions: Drug: IMVT-1401 (batoclimab)

INTERVENTIONS:
Drug: IMVT-1401 (batoclimab) — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody.
  Other Names: IMVT-1401

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 24 weeks of treatment with batoclimab in adult participants with biochemically documented hyperthyroidism due to GD who have failed to achieve euthyroidism on antithyroid drugs (ATDs).

ELIGIBILITY:
Inclusion Criteria:

* Have serologically confirmed GD as documented by presence of elevated stimulatory thyrotropin receptor antibody (TSH-R-Ab) level (i.e., > specimen-to-reference ratio of 140%) at the Screening Visit.
* Have active hyperthyroidism due to GD with the following laboratory values at the Screening Visit:

  * TSH < LLN
  * FT3 > upper limit of normal (ULN) and <=5 * ULN
  * FT4 > ULN and <=5 * ULN

Note: Participants who have T3 thyrotoxicosis (i.e TSH <LLN, FT3 > ULN and ≤5× ULN, but FT4 within normal range) at the Screening Visit may be enrolled, if they have serologically confirmed GD as per Inclusion Criterion 1.

* Are willing and capable of giving written informed consent, which includes being able to comply with all aspects of the study treatment and testing schedule.

Exclusion Criteria:

* History of hyperthyroidism not caused by GD (e.g., toxic adenoma or toxic multinodular goiter), and/or history or presence of thyroid storm.
* History of treatment with radioactive iodine or thyroid surgery.
* Total immunoglobulin G (IgG) level <6 grams per liter (g/L) at the Screening Visit.
* Albumin level <3.5 grams per deciliter (g/dL) (<35 g/L) at the Screening Visit.
* Absolute neutrophil count <1000 cells per cubic millimeter (cells/mm^3) at the Screening Visit.

Other, more specific exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who achieve normalization of free triiodothyronine (FT3) and free thyroxine (FT4), or have FT3 and/or FT4 below the lower limit of normal (LLN) at week 24 without increase in ATD dose | At Week 24

SECONDARY OUTCOMES:
Percentage of participants who achieve normalization of FT3 and FT4 at Week 24 with ATD dose <= 50% of the ATD dose at Week 24 | At Week 24
Percentage of participants who are off ATD treatment and achieve normalization of FT3 and FT4, or have FT3 and/or FT4 below the LLN at Week 24 | At Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Site Number - 6505, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No